CLINICAL TRIAL: NCT05410392
Title: Telemedicine Intervention in Patients With Chronic Pain in PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: N3769-R
Record Dates: First submitted 2022-06-02; First posted 2022-06-08 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Pain
MeSH Terms: conditions — Parkinson Disease; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Combined physical and cognitive exercise intervention (Experimental): Participants will receive both the physical exercise intervention and the cognitive exercise intervention for 3 months.
  Interventions: Behavioral: Physical exercise intervention; Behavioral: Cognitive exercise intervention
- Physical exercise intervention (Experimental): Participants will receive the physical exercise intervention for 3 months.
  Interventions: Behavioral: Physical exercise intervention
- Cognitive exercise intervention (Experimental): Participants will receive the cognitive exercise intervention for 3 months.
  Interventions: Behavioral: Cognitive exercise intervention
- Control group (Active Comparator): Participants will receive health education for 3 months.
  Interventions: Behavioral: Health education

INTERVENTIONS:
Behavioral: Physical exercise intervention — Home-based physical exercise with the use of a stationary recumbent style bike.
  Arms: Combined physical and cognitive exercise intervention; Physical exercise intervention
Behavioral: Cognitive exercise intervention — Home-based cognitive exercise with the use of smartphone to complete cognitive activities.
  Arms: Cognitive exercise intervention; Combined physical and cognitive exercise intervention
Behavioral: Health education — Provision of general information about a variety of topics
  Arms: Control group

SUMMARY:
Pain is a very common and disabling symptom in Parkinson's disease, yet it is often untreated. This study will assess the impact of home-based physical and cognitive exercise interventions to reduce pain in this disease. This approach would offer an easily implemented and affordable way to encourage and maintain use of these interventions by patients virtually indefinitely through remote access technology. The study findings may help VA clinicians provide optimal care for the many Veterans with Parkinson's disease and chronic pain.

DETAILED DESCRIPTION:
Project Background/Rationale: Pain is one of the most disabling and common nonmotor symptoms in Parkinson's disease (PD), with a prevalence of 40-85%. Research indicates that undertreatment of pain is particularly high in the PD population. Only about one-half of patients with PD who report pain receive regular pain medications. There is increasing interest in nonpharmacological treatments for chronic pain in PD to supplement pharmacological approaches. While there is evidence to support the utility of physical exercise to improve chronic pain management, relatively less is known about the role of cognitive exercise.

Project Objective: The investigators propose to conduct a pilot randomized, controlled trial in patients with chronic pain in PD to assess the impact of physical and cognitive exercise interventions on pain outcomes.

Project Methods: A total of 166 community-dwelling Veterans, 40 years of age or older, with chronic pain in mild-to-moderate PD will be randomly assigned in a 2 x 2 factorial design to one of four groups (1 - combined cognitive and physical intervention, 2 - physical intervention only, 3 - cognitive intervention only, 4 - health education). The investigators will test the effects of the interventions at 3 months for the outcome of pain severity.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of idiopathic PD
* At least 2 of the 3 cardinal signs of PD (resting tremor, rigidity, bradykinesia)
* Response to dopaminergic medication

Exclusion Criteria:

* Angina pectoris
* History of myocardial infarction (MI) within 6 months
* History of ventricular dysrhythmia requiring current therapy

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Pain Severity | 3 months
  Change in pain severity score from baseline to 3-month follow-up is the outcome

CONTACTS AND LOCATIONS:
Overall Officials: David William Sparrow, DSc, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No